CLINICAL TRIAL: NCT03236571
Title: Cardiorespiratory and Muscular Rehabilitation of Children and Young Adults With Marfan Syndrome: an Interventional, Prospective, Monocentric Study.
Brief Title: Cardiorespiratory and Muscular Rehabilitation of Children and Young Adults With Marfan Syndrome.
Acronym: Marfanpower
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/17/0257
Record Dates: First submitted 2017-07-28; First posted 2017-08-02 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2022-07

CONDITIONS: Marfan Syndrome
Keywords: Marfan syndrome; Personal Training Program; Cardiorespiratory rehabilitation; Muscular rehabilitation
MeSH Terms: conditions — Marfan Syndrome | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rehabilitation Program (Experimental): It will consist of 2 sessions of 40 minutes per week, for 12 weeks on ergometric bicycle. Each session of 40 min will include 5 minutes of warm-up, 5 minutes of recovery and 6 sequences of 5 min. Each 5-minute sequence will alternate between 4 minutes of pedaling at a load corresponding to the 1st ventilatory threshold (determined in the initial maximum cardiorespiratory effort test) and 1 minute of pedaling at a load corresponding to 2nd ventilatory threshold (determined in the initial maximum cardiopulmonary stress test).
  Interventions: Device: Rehabilitation program

INTERVENTIONS:
Device: Rehabilitation program — The rehabilitation program will consist of a Personalized Training Program and a muscle building program.

SUMMARY:
Marfan syndrome (MFS) is a rare genetic disease (1/5000) characterized by the association of ocular impairment, cardiovascular disease and musculoskeletal disease.

In some chronic conditions, physical activity and training have been shown to be effective in improving muscle strength and functional abilities but also fatigue and quality of life. We hypothesize that the implementation of a personalized exercise rehabilitation program (Personalized Training Program) in children and young adults with MFS, by improving muscle mass, physical endurance, muscle strength, bone mass and quality of life of these patients. In order to test this hypothesis, investigators wish to carry out an interventional, prospective, monocentric study for the first time in children and young adults (<25 years old) presenting an MFS.

DETAILED DESCRIPTION:
Marfan syndrome (MFS) is a rare genetic disease (1/5000) characterized by the association of ocular impairment, cardiovascular disease and musculoskeletal disease. Chronic fatigue and decreased physical endurance are almost constant complaints of patients with MFS (90% according to some studies), and have an impact on activities of daily living and quality of life. The fragility of the connective tissues and the muscle deficit, responsible for increased stress on the musculoskeletal system, may be involved in this symptomatology. This deficiency in muscle mass is already present in young children and worsens in adolescents and young adults, as researchers have shown in a clinical study carried out in the Toulouse MFS competence center. This muscle deficit may also explain, at least in part, the deficit in bone mass observed in children and adults.

In some chronic conditions, physical activity and training have been shown to be effective in improving muscle strength and functional abilities but also fatigue and quality of life. Investigators hypothesize that the implementation of a personalized exercise rehabilitation program (Personalized Training Program) in children and young adults with MFS, by improving muscle mass, physical endurance, muscle strength, bone mass and quality of life of these patients. In order to test this hypothesis, investigators wish to carry out an interventional, prospective, monocentric study for the first time in children and young adults (<25 years old) presenting an MFS.

ELIGIBILITY:
Inclusion Criteria:

* Marfan syndrome according to Ghent criteria.
* For minors, signed informed consent of at least one of the holders of the parental authority. For majors, signed informed consent.
* Patient affiliated to a social security scheme or equivalent.

Exclusion Criteria:

- Cardiac contraindications to Personal Training Program: O Severe aorta dilatation (aortic diameter> 45 mm) O and / or left ventricular failure (left ventricular ejection fraction <45%) O and / or severe mitral leakage ≥ grade 3

- Pregnancy

Ages: 7 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
Measurement of the maximum endurance capacities. | Month 9
  Reflected by the maximal oxygen consumption (VO2 peak) during an exercise test. The values of VO2 peak will be compared between the beginning and the end of the rehabilitation.

SECONDARY OUTCOMES:
Fatigability with effort and quality of life. | Month 9
  Questionnaires and self-assessment test. It will be compared between the beginning and the end of the rehabilitation.
Muscular force. | Month 9
  Static evaluation (handgrip) and dynamic evaluation by mechanography. It will be compared between the beginning and the end of the rehabilitation.
Body composition (muscle mass and bone mass). | Month 9
  Bone mineral content, bone mineral density of the entire body and lumbar spine (L2-L4), and muscle mass evaluated by dual-energy xray absorptiometry. It will be compared between the beginning and the end of the rehabilitation.
Aortic dilation and myocardial function. | Month 9
  Assessed by a cardiac ultrasound 2D and 2D strain. It will be compared between the beginning and the end of the rehabilitation.
Endothelial function. | Month 9
  Assessed by a high resolution vascular ultrasound. It will be compared between the beginning and the end of the rehabilitation.
Compliance. | Month 9
  Assessed by questionnaires. It will be compared between the beginning and the end of the rehabilitation.
Cardiac adverse events. | Month 9
  Evolution of the aorta dimensions, evaluated by ultrasound. It will be compared between the beginning and the end of the rehabilitation.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Edouard, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU de Toulouse, Toulouse, Midi-Pyrénées, France

REFERENCES:
- [Background] Judge DP, Dietz HC. Marfan's syndrome. Lancet. 2005 Dec 3;366(9501):1965-76. doi: 10.1016/S0140-6736(05)67789-6. PMID 16325700
- [Background] De Paepe A, Devereux RB, Dietz HC, Hennekam RC, Pyeritz RE. Revised diagnostic criteria for the Marfan syndrome. Am J Med Genet. 1996 Apr 24;62(4):417-26. doi: 10.1002/(SICI)1096-8628(19960424)62:43.0.CO;2-R. PMID 8723076
- [Background] Loeys BL, Dietz HC, Braverman AC, Callewaert BL, De Backer J, Devereux RB, Hilhorst-Hofstee Y, Jondeau G, Faivre L, Milewicz DM, Pyeritz RE, Sponseller PD, Wordsworth P, De Paepe AM. The revised Ghent nosology for the Marfan syndrome. J Med Genet. 2010 Jul;47(7):476-85. doi: 10.1136/jmg.2009.072785. PMID 20591885
- [Background] Bathen T, Velvin G, Rand-Hendriksen S, Robinson HS. Fatigue in adults with Marfan syndrome, occurrence and associations to pain and other factors. Am J Med Genet A. 2014 Aug;164A(8):1931-9. doi: 10.1002/ajmg.a.36574. Epub 2014 Apr 9. PMID 24719044
- [Background] Giske L, Stanghelle JK, Rand-Hendrikssen S, Strom V, Wilhelmsen JE, Roe C. Pulmonary function, working capacity and strength in young adults with Marfan syndrome. J Rehabil Med. 2003 Sep;35(5):221-8. doi: 10.1080/16501970306095. PMID 14582554
- [Background] Percheron G, Fayet G, Ningler T, Le Parc JM, Denot-Ledunois S, Leroy M, Raffestin B, Jondeau G. Muscle strength and body composition in adult women with Marfan syndrome. Rheumatology (Oxford). 2007 Jun;46(6):957-62. doi: 10.1093/rheumatology/kel450. Epub 2007 Feb 28. PMID 17329351
- [Background] Behan WM, Longman C, Petty RK, Comeglio P, Child AH, Boxer M, Foskett P, Harriman DG. Muscle fibrillin deficiency in Marfan's syndrome myopathy. J Neurol Neurosurg Psychiatry. 2003 May;74(5):633-8. doi: 10.1136/jnnp.74.5.633. PMID 12700307
- [Background] Haine E, Salles JP, Khau Van Kien P, Conte-Auriol F, Gennero I, Plancke A, Julia S, Dulac Y, Tauber M, Edouard T. Muscle and Bone Impairment in Children With Marfan Syndrome: Correlation With Age and FBN1 Genotype. J Bone Miner Res. 2015 Aug;30(8):1369-76. doi: 10.1002/jbmr.2471. Epub 2015 May 14. PMID 25656438
- [Background] Burks TN, Andres-Mateos E, Marx R, Mejias R, Van Erp C, Simmers JL, Walston JD, Ward CW, Cohn RD. Losartan restores skeletal muscle remodeling and protects against disuse atrophy in sarcopenia. Sci Transl Med. 2011 May 11;3(82):82ra37. doi: 10.1126/scitranslmed.3002227. PMID 21562229
- [Background] Peters KF, Horne R, Kong F, Francomano CA, Biesecker BB. Living with Marfan syndrome II. Medication adherence and physical activity modification. Clin Genet. 2001 Oct;60(4):283-92. doi: 10.1034/j.1399-0004.2001.600406.x. PMID 11683774
- [Result] Edouard T, Bajanca F, Flumian C, Marion-Latard F, Pradayrol C, Guitarte A, Langeois M, Van Kien PK, Yart A, Auriol F, Garrigue E, Dulac Y. A personalized home-based exercise training program in children with Marfan and Loeys-Dietz syndromes improves aerobic exercise capacity and health-related quality of life. Orphanet J Rare Dis. 2026 Feb 4. doi: 10.1186/s13023-026-04234-4. Online ahead of print. No abstract available. PMID 41639855
- [Derived] Edouard T, Picot MC, Bajanca F, Huguet H, Guitarte A, Langeois M, Chesneau B, Van Kien PK, Garrigue E, Dulac Y, Amedro P. Health-related quality of life in children and adolescents with Marfan syndrome or related disorders: a controlled cross-sectional study. Orphanet J Rare Dis. 2024 Apr 30;19(1):180. doi: 10.1186/s13023-024-03191-0. PMID 38685042